CLINICAL TRIAL: NCT02448394
Title: Assessment of a Community Support Worker Intervention for PLWH in Rural Ethiopia
Brief Title: Assessment of a Community Support Worker Intervention for Persons Living With HIV (PLWH) in Rural Ethiopia
Acronym: SHAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1410S54203
Record Dates: First submitted 2015-05-14; First posted 2015-05-19 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: HIV
Keywords: community support workers; retention in care

STUDY DESIGN:
Intervention Model Description: Randomized community trial
Who Masked: Investigator
Masking Description: Study investigators (except statistician and data manager) blinded to interim outcome results by study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): At each of the intervention sites, all newly enrolled participants will have an HIV community support worker (CSW) assigned them. Strong preference will be given to matching CSWs and clients from the same kebele (village or neighborhood of residence). CSW responsibilities include: education on HIV treatment and health promoting behaviors, social support/counseling, facilitated communication with the HIV clinic, referrals as needed for other support needs.
  Interventions: Other: Community Support Worker
- Standard of Care (No Intervention): At control sites, patients will receive standard of care facility-based medical care and counseling, consistent with general standards of care offered to HIV patients throughout the country as determined by the Ethiopian Ministry of Health.

INTERVENTIONS:
Other: Community Support Worker — At each of the intervention sites, all newly enrolled participants will have an HIV community support worker (CSW) assigned them. CSW responsibilities include: education on HIV treatment and health promoting behaviors, social support/counseling, facilitated communication with the HIV clinic, referrals as needed for other support needs.
  Arms: Intervention

SUMMARY:
This study, to be conducted in southern Ethiopia, is a randomized community trial, evaluating the use of local community support workers who provide for HIV patients education, counseling/social support, and linkage to the HIV Clinic. Patients will be followed for at least three years, with a primary goal of improving retention in HIV care, and secondary goals of improving client knowledge, attitudes about being HIV-positive, feelings of social support and clinical health status.

DETAILED DESCRIPTION:
As a critical gap in the HIV cascade of care in sub-Saharan Africa and elsewhere, many patients entering HIV care are lost to follow-up (LTFU), especially within the first 1-2 years. Many such patients die without treatment or return with advanced immune suppression. Our studies in Ethiopia indicate that HIV patients in rural settings (where HIV is increasingly treated) face multiple challenges that may impact retention in care and health status, including lack of knowledge about HIV treatment, internal and perceived stigma, social isolation, and poor access to the medical care system. Although HIV programs have used community support workers (CSWs) to address these and other challenges, evidence for efficacy of CSW programs is largely based on observational and single site studies, and factors associated with positive outcomes are not well understood.

During 2011-2012, we successfully implemented a pilot community intervention to support HIV patients in rural Ethiopia, using CSWs who were themselves HIV positive. Among HIV patients newly enrolled in care, LTFU was minimal, and clients had significant improvement in HIV knowledge, mental and physical quality of life, and perceived social support, with reduction in chronic symptoms and internal stigma.

Using an intervention grounded in the conceptual framework of social support as buffering against the negative effects of stressful events, we propose to rigorously evaluate a CSW intervention in a large multi-site community randomized trial. In Ethiopia's Southern Nations, Nationalities and Peoples' Region, 16 hospitals and 32 health centers will be randomized to intervention or control arms. For each intervention site, CSWs from that local area will be hired, trained, and assigned to HIV positive clients to provide in community settings: informational support (education/counseling); emotional support (to addressed internal and perceived stigma), companionship support (to reduce social isolation), and instrumental support (with increased access to the HIV clinical care system). 2,640 newly diagnosed HIV patients from these sites will receive a baseline assessment and will be followed for 36 months with yearly follow-up assessments with: (a) health surveys that include knowledge about HIV treatment, internal and perceived stigma, feelings of social support, and physical and mental health (quality of life), and (b) data from the clients' HIV Clinic record, including dates of clinic visits (to assess ongoing retention in care) clinical status, cluster of differentiation (CD4+) count and body mass index.

We hypothesize that compared to HIV patients in the control arm, those in the intervention arm will have reduced LTFU from HIV clinical care over 36 months of follow-up (Aim 1), and increased knowledge, feelings of social support, and health status, and decreased feelings of internal/perceived stigma and social isolation (Aim 2). We will also evaluate the extent to which factors in Aim 2 are predictive of retention in care (Aim 3). These results will have strong research implications to improve community programs to strengthen the HIV care continuum and decentralized HIV care not only in Ethiopia, but many other resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* new enrollment in HIV care at hospital or health clinic in the target region within the previous 3 months, and
* age >18 years

Exclusion Criteria:

* inability to give consent because of physical or mental incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1799 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Retention in care | 3-year follow-up
  Retention in HIV care will be defined as the fraction of all patients initiating care who continue to be alive and access HIV care (i.e., minus those who die, transfer to another care facility, or are lost to follow-up).

SECONDARY OUTCOMES:
Change in HIV knowledge | 3-year follow-up
  Knowledge will focus on HIV treatment-related issues
Change in HIV-related attitudes | 3-year follow-up
  Questions will be asked about a variety of attitudes, including those related to internalized HIV stigma and perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lifson, MD, Principal Investigator — University of Minnesota
Locations (5):
- Ethiopia (5):
  - Arba Minch Hospital, Arba Minch, Snnpr
  - Butajira Hospital, Butajīra, Snnpr
  - 29 Other Hospitals and Health Centers, Multiple Towns, Snnpr
  - Sodo Hospital, Sodo, Snnpr
  - National Alliance of State and Territorial AIDS Directors, Addis Ababa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lifson AR, Workneh S, Hailemichael A, MacLehose RF, Horvath KJ, Hilk R, Fabian L, Sites A, Shenie T. A multi-site community randomized trial of community health workers to provide counseling and support for patients newly entering HIV care in rural Ethiopia: study design and baseline implementation. HIV Clin Trials. 2018 Jun;19(3):112-119. doi: 10.1080/15284336.2018.1461999. Epub 2018 Apr 24. PMID 29688139